CLINICAL TRIAL: NCT03497208
Title: Comparative Study of Surgical Treatment of Vitiligo: Microneedling Versus Microneedling With Suspension of Uncultured Epidermal Cells
Brief Title: Comparative Study of Surgical Treatment of Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170596
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Vitiligo
Keywords: Surgery; melanocytes; dermarolling system
MeSH Terms: conditions — Vitiligo | interventions — Percutaneous Collagen Induction; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microneedling+cell susp+phototherapy (Experimental): Experiment is about the use of abrasion technic with dermaroller, equipped with a 0,25mm needle, applied on a vitiligo lesion. After that, a transplant with non cultured cell suspension (melanocytes and keratinocytes) will be applied to pacient 's skin scalp.
  Interventions: Procedure: Microneedling; Procedure: Cell suspension; Radiation: Phototherapy
- Microneedling and phototherapy (Active Comparator): Technique involves only the abrasion with dermaroller equipped with 0,25mm on the lesion of vitiligo.
  Interventions: Procedure: Cell suspension; Radiation: Phototherapy

INTERVENTIONS:
Procedure: Microneedling — The technique is about applying a dermaroller equipped with 0.25 mm needles over the vitiligo area.
  Arms: Microneedling+cell susp+phototherapy
Procedure: Cell suspension — The technique involves preparation of a cell suspension (keratinocyte/melanocyte) prepared by trypsinization from a non-lesioned part of a patient's scalp skin and transepidermal delivery using a dermarollerequipped with 0.25 mm needles.
Radiation: Phototherapy — The patient will receive phototherapy UVB-NB in the lesions of vitiligo after 15 days of the surgical procedure.

SUMMARY:
A comparative study for the surgical treatment of vitiligo in which the same patient will receive in acromic and symmetric lesions of vitiligo dermabrasion with micro needling and on the other side dermabrasion with micro needling followed by the application of cell suspension (melanocytes and uncultured keratinocytes). These cells will be removed from the own patient through the skin of the scalp. After the surgical procedure, patients will be submitted to UVB-NB phototherapy sessions (twice a week) and evaluated for repigmentation of vitiligo lesions at 14 and 24 weeks of treatment.

DETAILED DESCRIPTION:
Background: Vitiligo is characterized by a depigmentation acquired with partial or total loss of melanocytes from the epidermis, causing great psychosocial impact. Several therapeutic modalities have been proposed for its treatment and surgical treatments have been shown to be promising, especially in recalcitrant cases. The technique of epidermal rasping grafting, a variant of the punch micrografts technique, shows high repigmentation rates and does not require high cost technology. Objective: The objective of this project is to perform a comparative study for the surgical treatment of vitiligo, in which the same patient (N = 10) will receive, in symmetrical acrylic areas, only dermabrasion with a micro needling of 0.25 mm or dermabrasion using micro needling followed of the cell suspension application (melanocytes and uncultured keratinocytes). Methodology: In the donor area (scalp) the healthy tissue will be removed. This tissue will be placed in a sterile container with physiological saline and fragmented with delicate scissors for about 20 minutes until homogeneous consistency of the material is obtained. After the enzymatic digestion of epidermal cells of the dermis, it will isolate melanocytes and keratinocytes that will be placed in the recipient area. After 15 days of the surgical procedure, patients will start the phototherapy UVB-NB sessions (twice a week). The patients will be evaluated about the pain during the procedure, the improvement of injuries of vitiligo and the vitiligo-specific quality-of-life instrument (VitiQoL Vitqol Index) will be applied after and before the treatment. Conclusion: The technique of grafting by epidermal scrap shows high rates of repigmentation and does not require high cost technology, which motivated us, in this study, corroborating the literature and helping to disseminate this technique.

ELIGIBILITY:
Inclusion Criteria:

* Older than 14 years old
* Patients in treatment in the Dermatology Service HCPA
* Patients able to do UVB - NB phototherapy
* Patients with stable vitiligo lesions more than 1 year

Exclusion Criteria:

* Under 14 years old
* Patients unable to do phototherapy UVB-NB
* Unstable vitiligo lesions less than 1 year
* Patients with immunodeficiency (diabetes, infection, use of immunosuppressive drugs)
* Pregnancy and lactating
* Phototherapy session less than 2 months
* Patients with some kind of allergy about the drugs that will be used (like lidocaine anesthetic cream or chlorhexidine antiseptic)
* Patients using photosensitizing drugs
* Patients with keloids history, Hypertrophic scar or post inflammatory Hyperpigmentation.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-10-13 (Estimated); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
Evaluate the repigmentation of vitiligo lesion | The measure will be made in 24 weeks after the procedure
  Through a transparent millimeter paper the vitiligo area will be measure

SECONDARY OUTCOMES:
Vitiligo-specific quality-of-life instrument (VitiQoL). | 6 months
  A negative impact on vitiligo patients in terms of quality of life has been suggested. We propose evaluate the quality life in this patients after and before the treatment using the the vitiligo-specific quality-of-life instrument (VitiQoL).
Pain index | 6 months
  Evaluate in scale of 1 to 10 the pain of the procedure described by the patient
Index of satisfaction | 6 months
  Evaluate the satisfaction of the patient with this treatment using a scale of 1 to 5

CONTACTS AND LOCATIONS:
Overall Officials: Tania Cestari, Dr, Study Director — Federal University of Health Science of Porto Alegre
Locations (1):
- HCPA, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided